CLINICAL TRIAL: NCT03983265
Title: Condylar/Proximal Segments Repositioning Using CAD/CAM Generated Wafer After Bilateral Sagittal Split Osteotomy in Skeletal Mandibular Deformity
Brief Title: Condylar Segment Repositioning Using CAD/CAM Generated Wafer After BSSO in Skeletal Mandibular Deformity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yara mamdouh mustafa, Teaching Assistant, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ymmustafa
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Skeletal Abnormalities

STUDY DESIGN:
Intervention Model Description: Condylar/Proximal Segments Repositioning Using CAD/CAM Generated Wafer After Bilateral Sagittal Split Osteotomy in Skeletal Mandibular Deformity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- computer guided condylar reposition device (Other): surgical procedure : under general anesthesia after BSSO condyle will be repositioned by computer guided repostioning device
  Interventions: Other: Bilateral Sagittal Split Osteotomy

INTERVENTIONS:
Other: Bilateral Sagittal Split Osteotomy — after BSSO condyle will be re positioned by using computer guided device

SUMMARY:
Maintaining the condylar position after bilateral sagittal split ramus osteotomy (BSSO) is one of the most important aspects in terms of condylar function ,.An altered condylar position can cause internal derangement of the joint, loss of the mandibular angle, increased risk of relapse, condyle sagging, and impaired masticatory function.

In previous years, a great deal of attention has been paid to maintaining the preoperative condylar position during orthognathic surgery. Numerous condylar positioning methods have been reported and could be divided into manual/empirical methods, conventional methods , navigation, and sonographic monitoring, Computer guided methods which is more accurate than other methods

DETAILED DESCRIPTION:
unpredictable condylar position after orthognathic surgery, will lead to malocclusion, derangement of the condylar surface, condylar resorption, condylar sag, distraction of the condyles from the fosse. In previous years, several authors had been adopted several techniques to maintain the preoperative condylar position during orthognathic surgery. Numerous condylar positioning methods have been reported which could be divided into conventional techniques (manual maneuvers or aiding tools), Extra and intra oral navigational techniques , surgeons had been utilized these techniques in condylar repositiong after BSSO but it was time and effort consuming and sometimes it was inaccurate. the aim for conducting the research is accurate positioning of condyle three dimensionally to minimize effort and operating time of surgery .

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient above 18 years
* Patients needs bilateral sagittal split osteotomy
* All patients are free from any systemic disease that may affect normal bone healing
* Sufficient dentition to reproduce the occlusal relationships
* Patient's consent to participate

Exclusion Criteria:

* Patient with TMJ Disorders
* Patients with any systemic disease that may affect normal healing
* Intra-bony lesions or infections that may interfere with surgery.the presence of
* Previous orthognathic surgeries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of postoperative condylar position in relation to the corrected virtual model | immediate postoperative
  the accuracy of postoperative condylar position will be assessed using Mimics soft ware ,measuring unit (mm)

SECONDARY OUTCOMES:
operative time | during operation
  surgical time will be assessed via clinical assessment measuring unit (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed omara, Lecturer, Study Director — faculty of oral and dental medicine Cairo university
Locations (1):
- oral and dental medicine Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Computer-assisted orthognathic surgery: feasibility study using multiple CAD/CAM surgical splints — https://www.ncbi.nlm.nih.gov/pubmed/22668627
- See also: Orthognathic Positioning System: Intraoperative System to Transfer Virtual Surgical Plan to Operating Field During Orthognathic Surgery — https://www.ncbi.nlm.nih.gov/pubmed/23312847
- See also: Clinical and radiographic evaluation of a computer-generated guiding device in bilateral sagittal split osteotomies — https://www.ncbi.nlm.nih.gov/pubmed/24099655
- See also: A novel method for the management of proximal segment using computer assisted simulation surgery: correct condyle head positioning and better proximal segment placement — https://www.ncbi.nlm.nih.gov/pubmed/26258114